CLINICAL TRIAL: NCT03492567
Title: Study of Circulating Monocytes as Predictive Biomarker of Osteoclastogenesis in Cystic Fibrosis-related Bone Loss. Impact of CFTR Correctors.
Brief Title: Study of Circulating Blood Cell Monocytes as Predictive Biomarker of Bone Cystic Fibrosis Disease. Impact of CFTR Correctors.
Acronym: MUCO-OS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K171004J; 2017-A02965-48 (Other: ID-RCB)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; CFTR; CFTR modulators; Monocyte; Osteoclast; Osteoporosis
MeSH Terms: conditions — Cystic Fibrosis; Osteoporosis | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood monocyte precursors/osteoclasts (Experimental): Blood test
  Interventions: Biological: Blood test

INTERVENTIONS:
Biological: Blood test — Blood draw (max 15 ml)

SUMMARY:
The aim of the study is to look for risk factors of developing osteoporosis in patients with cystic fibrosis.

Blood cells called monocytes will be obtained from a blood sample. These monocytes will make possible to form another class of cells called osteoclasts in the laboratory. These latter cells are responsible for bone degradation and therefore promote the increase of bone fragility. The research will focus on the characterization of these cells to better understand their potential (low, medium or high) to increase bone fragility in patients with cystic fibrosis.

Finally the action of CFTR modulators on these bone cells will be tested.

DETAILED DESCRIPTION:
The aim of the study is to characterize the profile of circulating monocytes as predictive biomarker of osteoclastogenesis in CF related bone disease.

Investigators will evaluate the presence and regulation of CD115 (MCSF receptor) and CD265 (RANK) membrane receptors of circulating monocytes of cystic fibrosis patients.

They will also analyze the impact of the F508del CFTR mutation on the differentiation of monocytes into osteoclasts. We will 1) Quantify the training and functional activity of osteoclasts and, 2) Test in vitro the effects of correctors and potentiators of CFTR on the resorption activity of differentiated osteoclasts.

The study will be explained to patients and they only will have one blood test.

ELIGIBILITY:
Inclusion Criteria:

* patients with cystic fibrosis
* attending the Paris Cochin adult CF centre
* with at least F508del mutation (homozygote or heterozygote patients)

Exclusion Criteria:

* patients younger than 18
* absence of signed consent
* patients without a F508del mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Phenotype of CD14 monocytes/osteoclasts | 1 day

SECONDARY OUTCOMES:
In vitro test of CFTR modulators | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Dominique HUBERT, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, Paris, France

REFERENCES:
- [Result] Jourdain ML, Sergheraert J, Braux J, Guillaume C, Gangloff SC, Hubert D, Velard F, Jacquot J. Osteoclastogenesis and sphingosine-1-phosphate secretion from human osteoclast precursor monocytes are modulated by the cystic fibrosis transmembrane conductance regulator. Biochim Biophys Acta Mol Basis Dis. 2021 Mar 1;1867(3):166010. doi: 10.1016/j.bbadis.2020.166010. Epub 2020 Nov 11. PMID 33188942